CLINICAL TRIAL: NCT05920759
Title: Sex-specific Effect of Restricted Sleep on Brain Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jill Kanaley, Interim Chair & Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 2097207
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Cerebrovascular Circulation
MeSH Terms: interventions — Cerebrovascular Circulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Normal sleep (Placebo Comparator): Participants will sleep for 7-9 hours the night prior to the study visit.
  Interventions: Diagnostic Test: Cerebral blood flow
- Restricted sleep (Experimental): Participants will restrict sleep to four hours the night prior to the study visit.
  Interventions: Diagnostic Test: Cerebral blood flow

INTERVENTIONS:
Diagnostic Test: Cerebral blood flow — Transcranial Doppler (TCD) is a non-invasive diagnostic tool used to estimate cerebral blood flow velocity (CBFV), cerebral autoregulation, cerebrovascular reactivity (CVR), intracranial pressure, cerebral perfusion pressure as well as other indicators of cerebral hemodynamics and autoregulation.

SUMMARY:
The goal of this clinical trial is to compare the impact of restricted sleep on brain blood health in healthy men and women. The main question[s] it aims to answer are:

* Whether morning cerebral blood flow velocity is greater following a night of normal sleep compared to restricted sleep
* Whether the effect of sleep restriction on cerebral blood flow will be greater in males compared to females Participants will complete one 1-hour screening visit and two 2.5-hour study visits. Study visits will be conducted on two separate days.

DETAILED DESCRIPTION:
Transcranial Doppler (TCD) is a non-invasive diagnostic tool used to estimate cerebral blood flow velocity (CBFV), cerebral autoregulation, cerebrovascular reactivity (CVR), intracranial pressure, cerebral perfusion pressure as well as other indicators of cerebral hemodynamics and autoregulation. Whereas TCD has been widely used in research, clinical, and outpatient settings, studies specifically designed to examine the effect of limited sleep on brain health and potential impact of sex are sparse. Thus, the present study will investigate sex-specific differences in cerebral blood flow under conditions of normal and restricted sleep. Investigators will conduct measures of CBFV and CVR on two separate days under tightly controlled experimental conditions. This study hypothesizes greater morning cerebral blood flow velocity following a night of normal sleep compared to restricted sleep. This study further hypothesize the effect of sleep restriction on CBFV and CVR will be greater in males compared to females. Results from the present study will provide important data necessary to develop future, well-controlled studies examining the impact of long-term modifications in exercise and/or sleep on cerebral hemodynamics and, by extension, risk for cerebrovascular events (i.e. stroke).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women, 18-45 years of age, BMI 18-30 kg/m2, non-pregnant, non-breastfeeding, and non-nicotine users

Exclusion Criteria:

* any medications known to affect sleep, autonomic, metabolic, or cardiovascular health, have a self-reported history of hepatic, renal, pulmonary, cardiovascular, or neurological disease, stroke or neurovascular disease, bleeding/clotting disorders, sleep apnea or other sleep disorders, diabetes, history of alcoholism or substance abuse, major cardiovascular event or surgical procedure within the past three months, or hypertension

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow velocity | Two days
  Greater morning cerebral blood flow velocity following a night of normal sleep compared to restricted sleep

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States